CLINICAL TRIAL: NCT03941678
Title: The Effect of Creatine Supplementation and Resistance Training in Stroke Survivors
Brief Title: Creatine Supplementation During Resistance Training for People Recovering From Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Regina (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Parallel groups: creatine and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine (Experimental): 0.3 g/kg/d creatine for 7 days; 0.1 g/kg/d creatine for 63 days
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): 0.3 g/kg/d placebo for 7 days; 0.1 g/kg/d placebo for 63 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — 0.3 g/kg/day for 7 days; 0.1 g/kg/day for 63 days
  Arms: Creatine
Dietary Supplement: Placebo — 0.3 g/kg/day for 7 days; 0.1 g/kg/day for 63 days
  Arms: Placebo

SUMMARY:
Creatine monohydrate is important for sustaining phosphocreatine stores in tissues such as muscle and brain. Phosphocreatine is an important source of energy in these tissues. Supplementation with creatine monohydrate is effective in healthy and clinical populations for improving muscle and brain function. The purpose of our study is to determined whether creatine supplementation is effective during resistance training for improving muscle and brain function in people recovering from stroke.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of creatine supplementation and supervised resistance training in stroke survivors. It is hypothesized that creatine supplementation and resistance training will increase whole-body lean tissue mass, limb muscle thickness, muscle strength, tasks of functionality and cognition and decrease symptoms of depression and anxiety compared to placebo and resistance training.

Stroke is characterized by an abrupt disturbance in cerebral circulation causing a neurological deficit. It is a major cause of adult neurological disability in North America, often resulting in significant muscle loss, weakness and functional limitations. Disability associated with stroke limits independent living and social participation in at least half of all stroke survivors. A sedentary lifestyle after stroke can increase the risk for recurrent stroke, cardiovascular disease, and diabetes mellitus. All factors may adversely affect independence and quality of life. The majority of stroke survivors have residual impairments such as hemiparesis, spasticity, cognitive dysfunction, and aphasia, with full recovery reached in a small portion of these individuals. One of the major consequences of these impairments is physical inactivity which inevitably contributes to muscle loss, decreased muscle function (i.e. strength, endurance) and impaired functionality. One intervention which may help improve muscle mass, muscle function and functionality in stroke survivors is supervised resistance training. Resistance training does not lead to muscle spasticity in stroke survivors and has been shown to improve the ability to perform activities of daily living. Another intervention which may be beneficial for stroke survivors is creatine supplementation. Creatine has been shown to increase muscle mass, muscle function and tasks of functionality when combined with resistance training, possibly by influencing cellular hydration status, high-energy phosphate metabolism, muscle protein kinetics, satellite cells, anabolic growth factors, and inflammation. Creatine has also shown promise for improving cognition and symptoms of depression and anxiety; however, no study has examined the combined effects of creatine supplementation and resistance training in stroke survivors.

The study will be a double-blind, repeated measures design. In order to minimize group differences, participants will be matched according to age, gender, and type of stroke and then be randomized on a 1:1 basis to one of two groups, creatine monohydrate or placebo (corn-starch maltodextrin). Creatine and placebo will be similar in taste, color, texture and appearance. A research assistant will be responsible for randomization and another research assistant will prepare study kits. Each study kit will contain the participants supplement for the duration of the study, detailed supplementation instructions, as well as measuring spoons. For days 1-7, participants will ingest 0.3g/kg of creatine or placebo (0.075 g/kg x 4 times daily). This creatine dosing strategy has been shown to be effective for increasing intramuscular creatine stores. For subsequent days, participants will consume 0.1 g/kg/day of creatine or placebo as this creatine dosage is effective for increasing muscle mass. On training days, participants will consume their supplement within 5 minutes after each training session. On non-training days, supplements will be consumed at the participants leisure. Adherence with creatine supplementation, placebo, and resistance training will be assessed by training and supplementation compliance logs. A retrospective treatment identification will be administered to all participants upon completion of the study in order to assess whether participants thought they were administered creatine, placebo, or unsure about what supplement they consumed.

The dependent variables that will be measured at baseline and after the intervention include: (1) whole-body lean tissue mass (dual energy x-ray absorptiometry) (2) muscle thickness (elbow and knee flexors and extensors; ultrasonography), (3) muscle strength (1-repetition maximum leg press and chest press), (4) tasks of functionality (berg balance scale, 6-minute walk test) (5) cognition (Montreal Cognitive Assessment), (6) depression (The Center for Epidemiologic Studies- Depression Scale) and anxiety (Generalized Anxiety Disorder 7-item). Participants will also complete a 3-day food log at baseline and during the last week of supplementation and training to determine whether total calories consumed as well as macronutrient intake changed over the duration of the study. Participants will be instructed to record all food and beverages consumption during these 3 days. Food records will be analyzed using MyFitnessPal.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months post-stroke

Exclusion Criteria:

* creatine supplementation within the past 12 weeks
* medications affecting muscle function within the past 12 weeks
* kidney disorders
* liver disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Walking ability | Change from baseline to 10 weeks
  6-minute walk test (maximal distance)

SECONDARY OUTCOMES:
Lean tissue mass | Change from baseline to 10 weeks
  Lean tissue mass determined by DXA
Leg muscle thickness | Change from baseline to 10 weeks
  Knee extensor muscle thickness by ultrasound
Arm muscle thickness | Change from baseline to 10 weeks
  Biceps muscle thickness by ultrasound
Leg strength | Change from baseline to 10 weeks
  Leg press 1-repetition maximum
Upper body strength | Change from baseline to 10 weeks
  Chest press 1-repetition maximum
Balance | Change from baseline to 10 weeks
  Berg balance scale to measure balance. Includes 14 sub-scales which are summed. Scoring range is from 0 (worse) to 56 (best)
Cognition | Change from baseline to 10 weeks
  Montreal cognitive assessment to assess cognitive ability. Seven sub-scales which are summed. Scoring range is from 0 (worse) to 30 (best)
Anxiety | Change from baseline to 10 weeks
  General Anxiety Disorder Assessment to assess anxiety. Seven questions whose scores are summed. Scoring range is from 0 (least anxious) to 21 (most anxious)
Depression | Change from baseline to 10 weeks
  Center for Epidemiologic Depression (CES-D) Scale to assess depression. Twenty questions whose scores are summed. Scoring range is from 0 (least depressed) to 60 (most depressed)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Darren Candow, Ph.D., Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - Faculty of Kinesiology and Health Sciences, University of Regina, Regina, Saskatchewan
  - College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No